CLINICAL TRIAL: NCT05998889
Title: A Feasibility Study of a Combination of Graded Pain Exposure and Graded Motor Imagery in People With Complex Regional Pain Syndrome Type 1
Brief Title: Feasibility of a Combination of Graded Pain Exposure and Graded Motor Imagery in People With Complex Regional Pain Syndrome Type 1
Acronym: ABILITIES-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Principal Investigator, Jordi Alcaide Altet, Principal investigator, physiotherapist, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABILITIES-1
Record Dates: First submitted 2023-07-25; First posted 2023-08-21 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Complex Regional Pain Syndrome I (CRPS I)
Keywords: Complex Regional Pain Syndrome; Physiotherapy (specialty); Pain Management; Exposure Therapy; Efficacy; Safety
MeSH Terms: conditions — Complex Regional Pain Syndromes; Agnosia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: GPE+GMI (Experimental): Pain Education program based on Neuroscience of pain and the Fear-Avoidance model + Graded Pain Exposure Exercises + Graded Motor Imagery
  Interventions: Behavioral: Experimental group
- Control group: GMI (Active Comparator): Graded Motor Imagery
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Experimental group — Education, Graded Pain Exposure Exercises and Graded Motor Imagery. One supervision a week/9 weeks + exercises at home + encourage returning relevant activities despite pain
  Arms: Intervention group: GPE+GMI
Behavioral: Control group — Graded Motor Imagery following the GRaMI protocol, One supervision a week/9 weeks + exercises at home, activities encourage but pain contingency.
  Arms: Control group: GMI

SUMMARY:
Background:

There is low quality evidence supporting the use of rehabilitation in Complex Regional Pain Syndrome (CRPS), despite it is the first line approach in the Guidelines . Graded Motor Imagery (GMI) may be useful to improve pain and function at mid term (6 months). Graded Pain Exposure Approaches (GPE) seem to improve pain but not function at mid term. In other type of chronic pain conditions GPE offers better outcomes than "pain contingent" (exercises avoiding pain) approaches at short term (3 months) and similar at mid term. Following the recommendations of Authors, we will evaluate the efficacy and safety of a combined therapy of GMI and GPE in people with CRPS type 1.

Objective:

To evaluate the feasibility of a combined therapy of GPE and GMI in front of only GMI in people with CRPS-1 and the clinical impact on the primary outcome (Severity of the disease) of the intervention.

Design:

Feasibility Randomized controlled Trial, single blind of evaluator, 2 parallel arms. Measurement pre-intervention, post-intervention , 1 and 3 months follow-up.

Population:

People 18 years old or above with CRPS type 1 diagnosed by Budapest criteria and (1) without any psychological or psychiatric disease, (2) nor any neurosensorial issue that could compromise the realization of the therapy proposed (3) neither any major surgery intervention related to CRPS (e.g neurostimulation or sympathectomy) (4) nor minor intervention on the last 3 months (e.g. nerve blocks).

Outcomes:

Primary outcomes: Complex Regional Pain Syndrome Severity Scale (severity of the disease) and Safety Outcomes ( oedema, pain, temperature, Range of Motion). Secondary outcomes: 5Q-5D-5L (quality of life), SF-MPQ (Quality, Intensity and location of pain), PPT (pain pressure threshold), CPM ( pain inhibition pathways), FAAM or Quick Dash (function), PCS (catastrophism), Self efficacy in chronic pain questionnaire (self-efficacy), Dynamometry (Hand Grip strength),

ELIGIBILITY:
Inclusion Criteria:

* No difficulties understanding Spanish or Catalan.
* Diagnosed according to Budapest criteria.

Exclusion Criteria:

* Diagnosis of psychological or psychiatric illness
* Having received any major invasive treatment (e.g: Spinal cord Implants or sympathectomy of the affected extremity).
* Having received any minor invasive treatment (e.g: Nerves block) in the last three months.
* Having any neurosensorial difficulty that could compromise the execution of the therapy proposed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Severity of the disease | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Complex Regional Pain Syndrome Severity Score: This questionnaire contains self-reported items of persistent disproportionate pain, allodynia /hyperalgesia, asymmetry of temperature, color, sweating, oedema, trophic changes and motor changes . It also includes items observed by the examiner: allodynia , hyperalgesia , bilateral asymmetry of temperature by palpation, skin color changes, sweating, edema, trophic changes , and motor changes , as well as a decrease in active joint range of motion. The items are evaluated dichotomously; 0 indicates absence, and 1 indicates presence, resulting in a possible score range of 0 to 16, where higher scores indicate greater severity. The internal consistency obtained for the 16 items was adequate (Cronbach's α = 0.71).
Safety Outcome 1: oedema | Weekly during during the intervention (9 weeks)
  Perimetry ( measured with a measuring tape in centimeters ) of the metacarpofalangical joint line of the affected hand or the metatarsofalangical joint line of the affected foot. Control before and after the exercise intervention. Registered in a dichotomous way, absence if no changes observed, presence if the perimeter has raised 2 centimeters or more.
Safety Outcome 2: pain | Weekly during during the intervention (9 weeks)
  Changes in Verbal Pain Numerical Rating Scale after the exercises (recorded verbally). Control before and after the intervention. Registered in a dichotomous way, absence if no changes observed, presence if the Pain has raised 2 points or more.
Safety Outcome 3: temperature | Weekly during during the intervention (9 weeks)
  Changes in temperature (in Celsius Degrees, taken with a Hand Infrared thermometer). Control before and after the exercise intervention at 1 cm in the center of the back of the affected hand / foot and compared to the other side. Registered in a dichotomous way, absence if no changes observed, presence if the temperature raises 2ºC or more.
Safety outcome 4: range of motion | Weekly during during the intervention (9 weeks)
  Changes in active Range of Motion (measured with a finger goniometer in degrees). Control before and after the exercise intervention. Registered in a dichotomous way, absence if no changes observed, presence if active range of motion decreases 10º or more.

SECONDARY OUTCOMES:
Quality, Intensity and location of pain | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Mc-Gill Short Form Questionnaire : It is a self-administered questionnaire consisting of 15 descriptors, of which 11 are sensory categories and 4 are affective. Each pain descriptor contains four columns representing the categories 0: none, 1: mild, 2: moderate, and 3: severe. Participants must mark the level of descriptor that represents their pain. There is no cutoff score in the questionnaire; higher values indicate more pain. Additionally, the questionnaire includes a visual analog scale of pain, which is a validated and reliable metric for pain assessment
Pain pressure level | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Pain Pressure Threshold: Measured using a handheld pressure algometer (PAIN TEST™ FPX 50). Algometry has shown excellent interexaminer reliability (ICC 0.91). Pressure pain thresholds will be assessed on the dorsal side at 2 local points and one away from the hand; the local points are located at the proximal interphalangeal joint of the third finger (point 1) and at the space between the first and second metacarpals (point 2). Additionally, dorsally at the middle third of the forearm (point 3), the mean values of three consecutive measurements will be taken and compared to the contralateral side.
  For the lower extremity, two local points will be assessed on the foot and one at a distance; the local points are located at the metatarsophalangeal joint of the 1st (point 4) and 5th toes on the dorsal side of the foot (point 5), and the distant point is the Anterior Tibial Tuberosity of the same leg (point 6).
Conditioned Pain Modulation | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Cold Pressure Test; The experimental tonic pain will be induced by submerging the contralateral hand in cold water following the Cold Pressor Test (conditioning stimulus), and the assessment of pressure pain thresholds (test stimulus) will be performed before and during the application of the conditioning stimulus using a handheld algometer. The Cold Pressor Test (CPT) has shown to be a superior conditioning stimulus to pain by ischemia and is widely used to evaluate conditioned pain modulation. The CPT will involve keeping the contralateral hand submerged in water at 12±1ºC up to the wrist for a period of 2 minutes. The assessment of pressure pain thresholds will begin 45 seconds after immersion; the locations will be local to the affected extremity; for the upper extremity will be performed at point 2, and for the lower extremities at point 4.
Upper limb function | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Upper limb function will be analyzed using the Quick-Disabilities of the Arm, Shoulder, and Hand (QuickDASH) scale. This questionnaire consists of 11 items, with a minimum of 10 items needed to be validly completed. It assesses the difficulty in performing daily activities, work-related tasks, social or family relationships, as well as pain and difficulty sleeping on a Likert scale ranging from 1 (no difficulty/problem) to 5 (unable/extremely difficult pain). The average of the responses is calculated, subtracting 1 from the total, and then multiplied by 25 to obtain a percentage related to the degree of disability, where higher values indicate greater disability. The QuickDASH has shown excellent test-retest reliability assessed by Lin's concordance coefficient of 0.80 and internal consistency greater than 0.9.
Lower limb function | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Foot and Ankle Ability Measure: (FAAM) scale will be used. This 29-item questionnaire assesses the physical function of individuals with foot or ankle-related disabilities. It consists of two subscales: the first one with 21 items evaluates activities of daily living (ADLs), and the second one with 8 items assesses sports activities. Higher scores indicate better function. Each item is scored on a 5-point Likert scale ranging from 0 (unable to perform) to 4 (no difficulty), with the option to answer N/A (not applicable) in case the activity is limited by any other aspect not related to the foot or ankle. The FAAM scale demonstrates high internal consistency (Cronbach's α for ADLs 0.97 and for sports 0.93) and test-retest reliability for ADLs (ICC=0.90) and for sports (ICC=0.76)
Quality of life (EQ-5D-5L) | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  EQ-5D-5L questionnaire: The EuroQoL 5 dimensions 5 levels questionnaire assesses quality of life through five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L has demonstrated efficacy, reliability, and discriminative ability in multiple pathologies and populations. Users evaluate their perception of each dimension at the moment of assessment and have five Likert-type options ranging from 1 ("no problems") to 5 ("extreme problems"). The questionnaire also includes a Visual Analog Scale (VAS) for perceived quality of life. The set of values is categorized into a 5-digit code. The VAS is marked with a cross, and it indicates the perceived health status on that particular day.
Catastrophism | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Pain Catastrophizing Scale (PCS). The PCS is a self-administered questionnaire that assesses the construct of "Pain Catastrophizing" in response to the modulation of painful stimuli. It consists of 13 items that assess three different dimensions: rumination (items 8, 9, 10, 11), magnification (items 6, 7, 13), and helplessness (items 1, 2, 3, 4, 5, 12). The PCS shows reliable test-retest parameters (0.79) and internal consistency (Cronbach's α of 0.84)
Self-efficacy | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Self-efficacy in Chronic Pain Questionnaire: this questionnaire assesses three dimensions with 22 items: self-efficacy in symptom control (items 1-8), self-efficacy in physical functioning (items 9-17), and self-efficacy in pain management (items 18-22). Each question is scored from 0 ("not at all capable") to 10 ("completely capable"), with a range of values from 0 to 100. The questionnaire has a test-retest reliability of r=0.75 and internal consistency (Cronbach's α of 0.91).
Strength | Pre-treatment, post-treatment (9 weeks) and at 1 and 3 months follow-up after treatment.
  Hand-grip strength measured with a dynamometer: isometric handgrip strength will be calculated on the affected side using a JAMAR hydraulic dynamometer, while seated with a straight back and feet touching the ground. The elbow is flexed at a 90° angle, in a neutral position of forearm pronation and supination, close to the body, with a neutral wrist position, and in the most comfortable device position for the user (42). The user will be instructed to squeeze the device as hard as possible upon verbal command. Three measurements will be taken with 5 seconds of rest between each. The test-retest reliability of the handgrip strength measurement with this dynamometer is very high (r=0.88-0.93)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Alcaide Altet, PT, Principal Investigator — University of Vic - UCC
Locations (1):
- CAP El Maresme, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shafiee E, MacDermid J, Packham T, Walton D, Grewal R, Farzad M. The Effectiveness of Rehabilitation Interventions on Pain and Disability for Complex Regional Pain Syndrome: A Systematic Review and Meta-analysis. Clin J Pain. 2023 Feb 1;39(2):91-105. doi: 10.1097/AJP.0000000000001089. PMID 36650605
- [Background] Harden RN, McCabe CS, Goebel A, Massey M, Suvar T, Grieve S, Bruehl S. Complex Regional Pain Syndrome: Practical Diagnostic and Treatment Guidelines, 5th Edition. Pain Med. 2022 Jun 10;23(Suppl 1):S1-S53. doi: 10.1093/pm/pnac046. PMID 35687369
- [Background] Smart KM, Ferraro MC, Wand BM, O'Connell NE. Physiotherapy for pain and disability in adults with complex regional pain syndrome (CRPS) types I and II. Cochrane Database Syst Rev. 2022 May 17;5(5):CD010853. doi: 10.1002/14651858.CD010853.pub3. PMID 35579382
- [Background] Smith BE, Hendrick P, Smith TO, Bateman M, Moffatt F, Rathleff MS, Selfe J, Logan P. Should exercises be painful in the management of chronic musculoskeletal pain? A systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(23):1679-1687. doi: 10.1136/bjsports-2016-097383. Epub 2017 Jun 8. PMID 28596288
- [Background] van de Meent H, Oerlemans M, Bruggeman A, Klomp F, van Dongen R, Oostendorp R, Frolke JP. Safety of "pain exposure" physical therapy in patients with complex regional pain syndrome type 1. Pain. 2011 Jun;152(6):1431-1438. doi: 10.1016/j.pain.2011.02.032. Epub 2011 Apr 6. PMID 21474244